CLINICAL TRIAL: NCT00553137
Title: Oral Candidiasis in HIV Infected Individuals in Tanzania
Brief Title: Single Dose Versus Two Weeks Course of Fluconazole in the Treatment of Oropharyngeal Candidiasis in HIV Infected Individuals in Tanzania
Acronym: SDVS2WK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Netherlands Organisation for Scientific Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fluc trial tz
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Oropharyngeal Candidiasis
Keywords: oropharyngeal candidiasis
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): single dose fluconazole (750 mg) and placebos 150 mg tablets once daily for 14 days
  Interventions: Drug: fluconazole
- 2 (Active Comparator): 150 mg fluconazole once daily for 14 days and placebos (5 placebos tablets) 750 mg once
  Interventions: Drug: fluconazole

INTERVENTIONS:
Drug: fluconazole — 750 mg (5 tablets of 150 mg tablets)taken once
  Arms: 1
Drug: fluconazole — 150 mg fluconazole tablets once daily for 14 days
  Arms: 2

SUMMARY:
A prospective randomized double blinded placebo controlled comparative trial will be performed at HIV clinic of the Muhimbili National Hospital/MUCHS where 220 HIV positive patients presenting with oropharyngeal candidiasis (OPC) on antiretroviral (ARVs) treatment or not will be included.

The aim of this study is to compare the efficacy and safety of single dose fluconazole (750mg) and two weeks course of fluconazole (150mg once daily)in the treatment of OPC in HIV positive patients. It is hypothesised that the two regimens are equally effective in the treatment of OPC.

DETAILED DESCRIPTION:
A structured standard questionnaire will be used to systematically collect essential data including demography, treatment history and concomitant infections and treatment.

General and oral examination, collection of oral isolates, mycological, hematological and biochemical investigations will be done at baseline and at end of treatment day 13-14.

All Patients will be followed up to 30 days after end of treatment for relapse

ELIGIBILITY:
Inclusion Criteria:

* HIV infection (as determined by positive ELISA and confirmed by Western blot)
* 18 years of age and above
* clinical picture of OPC, characterized by creamy, white, curd like patches, removable by scraping or by typical erythematous lesions (smooth red patches) on the oral mucosa, hard or soft palate and/or dorsal surface of the tongue; and microbiologically by visualization of yeast cells in Potassium hydroxide (10% KOH) preparations prepared from swab of visible lesions and confirmed positive Candida species culture

Exclusion Criteria:

* Patients who are currently receiving antifungal therapy or who had received such treatment within three days prior to enrollment in this study
* History of allergy to azole derivatives
* Abnormal liver function tests defined as alanine aminotransferase (ALT), aspartate aminotransferases (AST), or total bilirubin greater than three times the upper limit of normal; or clinical evidence of significant hepatic or renal disease within two months prior to enrollment
* Inability to tolerate oral drug administration; pregnancy or breast feeding; life expectancy of less than four weeks
* Participation in another drug study at the time of enrollment, treatment with drug which interact with fluconazole, such as vitamin K antagonists, warfarin, sulfonylurea anti-diabetic agents, rifampicin, phenytoin, isoniazid, carbamazepine and cisapride
* Documented systemic fungal infections, symptoms suggestive of esophageal candidiasis such as retrosternal chest pain, dysphagia or odynophagia unless this condition has been ruled out by endoscopic examination.
* Patients with history of alcohol abuse, drug addiction and psychiatric disorder, inability to cooperate and poor motivation will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
clinical and mycological cure | two weeks

SECONDARY OUTCOMES:
recurrence post treatment | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omar JM Hamza, DDS, Principal Investigator — Department of Oral Surgery and Oral Pathology, Muhimbili University College of Health Sciences; Mecky IN Matee, PhD, Study Chair — Department of microbiology, Muhimbili University College of Health Sciences; Ferdinand Mugusi, MD,MMED, Study Chair — Department of Internal Medicine, Muhimbili University College of Health Sciences; Andre JA Van der Ven, PhD, Study Director — Centre for Infectious Disease, Internal Medicine Department, Radboud University Nijmegen, the Netherlands; Paul E Verweij, PhD, Study Chair — Department of Medical Microbiology, Radboud University Nijmegen, the Netherlands
Locations (1):
- ART clinic Muhimbili National Hospital/Muhimbili University College of Health Sciences, Dar es Salaam, Dar es Salaam Region, Tanzania

REFERENCES:
- [Derived] Hamza OJ, Matee MI, Bruggemann RJ, Moshi MJ, Simon EN, Mugusi F, Mikx FH, van der Lee HA, Verweij PE, van der Ven AJ. Single-dose fluconazole versus standard 2-week therapy for oropharyngeal candidiasis in HIV-infected patients: a randomized, double-blind, double-dummy trial. Clin Infect Dis. 2008 Nov 15;47(10):1270-6. doi: 10.1086/592578. PMID 18840077